CLINICAL TRIAL: NCT06990360
Title: Accuracy of Computer Guided Implant Placement in Edentulous Mandible A Three-Dimensional In Vitro Study
Status: Completed | Type: Observational
Sponsor: Eslam Nashaat Saied Ahmed Mohamed (Other)
Responsible Party: Sponsor-Investigator, Eslam Nashaat Saied Ahmed Mohamed, Post graduate student, Future University in Egypt
Organization: Future University in Egypt (Other)
Other Study IDs: FUE.REC (13)/12-2017; Future University (Other: Future University)
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Edentulous Alveolar Ridge; Edentulous Alveolar Ridge In Mandible
Keywords: Computer-guided implant placement; Edentulous mandible; 3D printed surgical guide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBCT Scanning — The Styrofoam mandibles were scanned using CBCT, which was performed for each mandible pre-operatively, the raw DICOM data set obtained from the CBCT scanning were imported to a special third-party software* for secondary reconstruction.

SUMMARY:
Five stryofoam mandibles were included in this study to assess the accuracy of using computer guided surgical stent in placement of dental implants. The mandibles were CBCT scanned and imported to 3diagnosys software to implant planning. 8 implants were placed in each mandible virtually, 4 anterior implants and 4 posterior implants were placed. The plan was exported as STL file to be imported to the CAD software for designing of the stent. The surgical stent is printed using Micro DGP printer and invision tec e-shell 600 clear resin was used. Stainless steel sleeves were placed in the surgical guide then placed in ethanol 99% to remove the excess monomer.

The stent in placed over the mandible and sequential drilling was done until the desired osteotomies width was approached followed by the placement of the implants. Post-operative CBCT was done for the mandible including the implants to assess the accuracy, angulation and position of the placed implants

ELIGIBILITY:
Inclusion Criteria:

* Five styrofoam mandibles

Exclusion Criteria:

* no fractures or pathology

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Five styrofoam mandibles
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Mesiodistal (MD) Angle | 1 year
  measures in the software in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- future university in Egypt, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol